CLINICAL TRIAL: NCT06006351
Title: Comparison of the Effects of Exercise and Hypervolt Device Application on Pain, Muscle Strength and Normal Joint Movement in the Treatment of Shoulder Impingement Syndrome
Brief Title: Efficiency of Hypervolt Device Application in the Treatment of Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar54
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Exercise therapy and Applying a Hypervolt massager
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): classical physiotherapy protocol will be applied.
  Interventions: Other: Physiotherapy
- Massage (Experimental): In addition to the classical physiotherapy protocol, a Hypervolt Device will be applied.
  Interventions: Other: Physiotherapy; Other: Hypervolt Device

INTERVENTIONS:
Other: Physiotherapy — manual therapy stretching exercises strengthening exercises electrotherapy applications
Other: Hypervolt Device — The painful area will be applied with a massage tool, and the frequency and mode of the tool will be adjusted in a way that does not disturb the patient.
  Arms: Massage

SUMMARY:
The aim of this study is to compare the effects of exercise and Hypervolt Device on pain, muscle strength and normal joint movement in the treatment of shoulder impingement syndrome.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. The study sample will be divided into two groups by simple randomization method. Only exercise will be applied to 30 individuals diagnosed with shoulder impingement in the first group of the study. In the second group, 30 individuals with shoulder impingement diagnosis will be given a Hypervolt Device in addition to the exercise. Disabilities of the Arm, Shoulder and Hand Questionnaire, Visual Analog Scale and Lawton Daily Living Activities Questionnaire will be applied to the participants before and after the treatment. The obtained data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-50.
* Having a Visual Analogue Scale (VAS) value of 5 or higher.
* Having a history of shoulder pain for at least 1 month.
* Volunteer to participate in research.
* Having been diagnosed with Shoulder Impingement.

Exclusion Criteria:

* Having cognitive, mental or psychological problems.
* Having a condition that prevents him from exercising.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Questionnaire | 12 weeks
  It was developed to evaluate functional status and symptoms by focusing on physical function in upper extremity injuries. According to the results of the survey; a result from 0-100 is obtained from each part; 0-no apology 100-maximum apology.
Lawton Activities of Daily Living Scale | 12 weeks
  It is a questionnaire consisting of eight questions, including information about using the telephone, preparing food, shopping, doing daily household chores, washing clothes, getting on a transportation vehicle, using medicines and managing money. If the individual does the activities independently, three points, two points if he does it with help, and one point if he cannot do it at all. In Lawton Activities of Daily Living Scale; 0-8 points are classified as "dependent", 9-16 points as "semi-dependent", 17-24 points as "independent".

CONTACTS AND LOCATIONS:
Overall Officials: Tuba KARACA, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Consigliere P, Haddo O, Levy O, Sforza G. Subacromial impingement syndrome: management challenges. Orthop Res Rev. 2018 Oct 23;10:83-91. doi: 10.2147/ORR.S157864. eCollection 2018. PMID 30774463
- [Background] Ellenbecker TS, Cools A. Rehabilitation of shoulder impingement syndrome and rotator cuff injuries: an evidence-based review. Br J Sports Med. 2010 Apr;44(5):319-27. doi: 10.1136/bjsm.2009.058875. PMID 20371557
- [Background] Marik TL, Roll SC. Effectiveness of Occupational Therapy Interventions for Musculoskeletal Shoulder Conditions: A Systematic Review. Am J Occup Ther. 2017 Jan/Feb;71(1):7101180020p1-7101180020p11. doi: 10.5014/ajot.2017.023127. PMID 28027039
- [Background] Gebremariam L, Hay EM, van der Sande R, Rinkel WD, Koes BW, Huisstede BM. Subacromial impingement syndrome--effectiveness of physiotherapy and manual therapy. Br J Sports Med. 2014 Aug;48(16):1202-8. doi: 10.1136/bjsports-2012-091802. Epub 2013 Nov 11. PMID 24217037
- [Background] Steuri R, Sattelmayer M, Elsig S, Kolly C, Tal A, Taeymans J, Hilfiker R. Effectiveness of conservative interventions including exercise, manual therapy and medical management in adults with shoulder impingement: a systematic review and meta-analysis of RCTs. Br J Sports Med. 2017 Sep;51(18):1340-1347. doi: 10.1136/bjsports-2016-096515. Epub 2017 Jun 19. PMID 28630217